CLINICAL TRIAL: NCT01400685
Title: Lenalidomide in Combination With Bendamustine and Rituximab for Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma(CLL/SLL): a Phase I Study
Brief Title: Lenalidomide Plus Bendamustine and Rituximab for Untreated CLL/SLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-016
Record Dates: First submitted 2011-04-11; First posted 2011-07-22 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; B Chronic Lymphocytic Leukemia
Keywords: CLL; Leukemia; Untreated; B-CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Leukemia | interventions — Lenalidomide; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide will be dose escalated until the maximum tolerated dose is reached. The starting dose is 2.5mg, followed by 5mg, followed by 10mg.
  Other Names: CC-5013; Revlimid
Drug: Bendamustine — 90 mg/m^2 IV days 1-2 of each cycle for 6 cycles
  Other Names: Treanda; SDX 105
Drug: Rituximab — 375 mg/m^2 IV day 1 (cycle 1), 500 mg/m^2 day 1 (cycles 2-6)
  Other Names: Rituxan; Mabthera

SUMMARY:
Lenalidomide belongs to a group of drugs called immunomodulatory drugs (IMiD) that can modify or regulate the functioning of the immune system. It is an FDA approved drug for people with multiple myeloma. It is not currently approved for use in Chronic Lymphocytic Leukemia (CLL), but it does appear effective in CLL when used alone, and is being studied for use in combination with chemotherapy in this and other lymphomas and leukemias.

In this research study we are hoping to learn more about the effects of lenalidomide on CLL when given in combination with bendamustine and rituximab, which is a highly effective regimen for initial therapy of CLL/SLL. The investigators will be looking for the highest dose of lenalidomide that can be given safely, without causing any serious or unmanageable side effects.

DETAILED DESCRIPTION:
Subjects will receive lenalidomide, bendamustine and rituximab in cycles of 28 days (4 weeks). Lenalidomide will be administered orally once daily on days 8-21 of cycle 1 and on days 1-21 of all subsequent cycles. Bendamustine will be administered through a vein (IV infusion) on days 1 and 2 of each cycle. Rituximab will be administered as an IV infusion on day 1 of each cycle.

Subjects will receive routine blood tests and physical exam during each cycle. Tumor assessments by CT scan will be performed during cycles 2, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with B-cell CLL or SLL (chronic lymphocytic leukemia or small lymphocytic leukemia)
* Life expectancy > 3 months
* Organ and marrow function with protocol parameters
* Able to take aspirin daily

Exclusion Criteria:

* Age >80 years
* Prior systemic therapy for CLL/SLL including chemotherapy or antibody therapy
* Pregnant or breast-feeding
* Serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing informed consent
* Known hypersensitivity to thalidomide or lenalidomide
* Prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* HIV positive
* Prior history of another malignancy unless disease free for at least 2 years
* Uncontrolled intercurrent illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Identify the maximum tolerated dose of lenalidomide when combined with bendamustine and rituximab in CLL/SLL | 2 years

SECONDARY OUTCOMES:
Define dose limiting toxicities of bendamustine, rituximab and lenalidomide in CLL | 2 year
Clinical efficacy | 2 years
  response rate, progression-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, M.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts